CLINICAL TRIAL: NCT06624904
Title: The Effects of Single-dose Losartan on Social Processing in Healthy Adults: a Randomized Controlled Study
Brief Title: Losartan and Social Processing
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Oxford Health Biomedical Research Centre (OH BRC) support scheme (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: R92661
Record Dates: First submitted 2024-09-23; First posted 2024-10-03 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2024-09

CONDITIONS: Social Cognition
Keywords: Social Processing; Losartan; Renin Angiotensin System
MeSH Terms: interventions — Losartan

STUDY DESIGN:
Intervention Model Description: Parallel randomised experimental medicine trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Losartan (Experimental): 50 mg single-dose losartan
  Interventions: Drug: Losartan potassium 50mg
- Placebo (Placebo Comparator): Microcellulose placebo in identical capsule
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Losartan potassium 50mg — Single dose losartan (50 mg), encapsulated identically to placebo.
  Other Names: Losartan; Cozaar
  Arms: Losartan
Other: Placebo — Single tablet encapsulated identically to placebo.
  Arms: Placebo

SUMMARY:
This study explores the effects of single-dose losartan (50mg) versus placebo on social processing in healthy volunteers.

DETAILED DESCRIPTION:
While renin-angiotensin mechanisms have been implicated in physiological disease, such as hypertension and stroke, the discovery of a local brain renin-angiotensin system (RAS) in the 1970s brought into question whether the RAS may play a role in psychiatric disorders too. Recent work has supported this link, with several studies reporting RAS influence on aversive learning, stress response to traumatic stimuli, and fear extinction.

Despite these promising results, studies have yet to fully explore the influence of the RAS and losartan on social processes. It is plausible that the RAS may be involved in social functioning, as recent work reported that losartan reduces sensitivity to social punishment in healthy volunteers. Such an effect of losartan may have broad relevance for psychopathology, as impairment to social functioning is present across a range of psychiatric disorders.

In this double-blind, randomized between-group study, the investigators will examine the effects of a single dose of losartan (50mg) versus placebo on social processing in N=68 healthy volunteers. Following a one-hour waiting period, participants will complete a set of computer tasks investigating social processes reported to be sensitive to psychopathology. Specifically, participants will complete the Approach Avoidance Task which assesses social approach and avoidance behaviour in response to various facial expressions via joystick movement, the Interpretation Inflexibility Task which evaluates cognitive flexibility in a social context, the Social Learning Trust Game which evaluates social learning through a trust game between participant investors and realistic trustees, and Cyberball, which probes response to social rejection. Results from this study will provide more insight on the potential role of the RAS in social cognitive processing in humans, which could lead to an improved mechanistic understanding of emotional disorders that are marked by social impairment.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Aged 18-50 years
* Sufficient written and spoken English skills to understand what the study involves, and to complete the questionnaires
* Non- or light-smoker (5 cigarettes a day, if vaping: less than 50 puffs)
* BMI between 18 - 30

Exclusion Criteria:

* Current DSM-5 axis-I diagnosis (based on SCID results at screening) or history of a severe psychological disorder such as psychotic disorder, bipolar disorder, alcohol or substance abuse, or post-traumatic stress disorder
* First-degree family member with severe psychiatric illness (including psychosis, bipolar disorder, unipolar psychotic depression).
* CNS-medication last 6 weeks (including as part of another study)
* Current blood pressure or other heart medication, including aliskiren and beta blockers)
* Diagnosis of intravascular fluid depletion or dehydration
* History of angioedema
* Impaired kidney function (based on self-report)
* Very low blood pressure (defined as repeated (at least three consecutive measurements) measures of blood pressure under standardised conditions where either the systolic or the diastolic blood pressure or both are below 90/50 mmHg (in accordance with established standard definitions)
* Lifetime history of epilepsy or other neurological disorder, as established by a professional diagnosis (e.g. autism, ADHD)
* Lifetime history of systemic infection, or clinically significant hepatic, cardiac, obstructive respiratory, renal, cerebrovascular, metabolic, endocrine or pulmonary disease or disorder which, in the opinion of the investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study
* Significant loss of hearing that is not corrected with a hearing device
* Women: pregnancy (as determined by a urine test, if the participant's pregnancy status is unknown during the in-person visit), breast-feeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
AAT effect score | 1 hour after capsule intake
  mean reaction time of the pull trials of a valence category subtracted from the push trials of the same category, yielding a single indicator of approach/avoidance, with positive scores indicating relatively stronger approach and negative scores indicating relatively stronger avoidance

SECONDARY OUTCOMES:
Sensitivity to Social Rejection | 1 hour after capsule intake
  a) feelings of belonging, control, self-esteem, meaningful existence (on a scale from 1 to 5, with some items reverse coded) as measured on the reflexive and reflective needs-threat scale following Cyberball.
Social Learning | 1 hour after capsule intake
  Social learning rate (early round versus late round investment decisions by generosity condition)
Interpretation Inflexibility | 1 hour after capsule intake
  Within-person revision of biased interpretations: calculated by taking the average of differences between bias scores between stage 3/2 and 2/1. These two differences will be squared before averaging to reflect absolute change (i.e., in either direction), then the square root of the resulting average will be taken. Higher values mean more flexibility in revising prior interpretations.

CONTACTS AND LOCATIONS:
Locations (1):
- Warneford Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided